CLINICAL TRIAL: NCT01876277
Title: What Are the Psychosocial Implications of Body Image Issues in Adolescent Males With Cancer?
Brief Title: Body Image Issues in Boys Being Treated at the Royal Marsden
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 890-PSY-13; CCR3985 (Other: Royal Marsden NHS Foundation Trust)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: Cancer; Body image; Adolescent
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescent males with cancer: Males aged 13-21 who have been treated at the Royal Marsden Hospital for cancer.

SUMMARY:
In adolescence, the effects of cancer and its treatment can lead to bodily changes such as hair loss, weight loss or gain, amputations, scars and developmental delay. As treatments for childhood cancers improve and life expectancy increases, more adolescents have to deal with the effects of cancer and the treatment on their bodies throughout their lives.

Body image can be defined as "The mental image we hold of our bodies". There are two aspects to this, how we "see" our size/shape/weight etc, and then how we feel about this. Often the actual change in body does not always predict how people cope with it, or how they feel about it.

Prior research suggests, and clinical experiences suggests that body image issues arise for at least some adolescents with cancer, however it is unknown whether a disturbance in body image is seen as distressing for the adolescent, or how this affects them psychologically.

Body image problems were always seen as a typically female problem, and therefore researchers have often neglected to look at the issues for men. There is currently no research specifically addressing the impact of body image in adolescent boys with cancer.

This research will involve interviewing adolescent males with cancer with the aims to find out;

1. What the body image issues are, if any for this group.
2. How any body image issues might affect them, particularly psychologically.
3. What helps or hinders this group maintain a positive body image, or stop it having a negative impact on them psychologically.

It is hoped that this will help to inform psychological treatments for body image difficulties in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Male- as this research has identified a need for research with this particular group.
2. Aged between 13 and 21 (inclusive)as this research is focussing on adolescents and we have defined the age range of adolescence as 13 to 21, in line with other research on adolescence.
3. Have a diagnosis of cancer (any type)as this study is not focussing on any particular type of cancer and this will ensure a sufficient pool of participants.
4. Have been diagnosed for at least 6 months as issues about adjusting to the diagnosis will be less prevalent at this time and they are likely to have received some treatment for cancer which often produces some of the bodily changes that may affect their body image.
5. Have a prognosis of more than 3 months, as it would be unethical to interview people in the final stages of terminal cancer as end of life issues would be more prevalent. Three months was decided upon because often this is the length of time given to patients when it is decided that treatment is no longer indicated and their illness is considered terminal. We would not contact anyone whose cancer was considered terminal.
6. Have had treatment within the past 5 years, because beyond this time they are less likely to have body image issues and other issues or than cancer could be more prevalent for them, so they are not suitable participants.
7. Able to participate in the interview verbally and in English because the qualitative method requires detailed analysis of the texts and translation may lead to a loss in some of the meaning that is crucial for this research.

Exclusion Criteria:

* Any participant who did not meet all of the inclusion criteria would be excluded.

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent males who have been treated for cancer at the Royal Marsden Hospital within the past 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Qualitative Interview Schedule | 1 hour
  Interview schedule developed by researcher to act as topic guide for interview.

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Christopher, BSc, Principal Investigator — University of Surrey
Locations (1):
- Royal Marsden Hopstial, Sutton, London, United Kingdom